CLINICAL TRIAL: NCT03537976
Title: Targeting Surgeons' Decision-Making for Cleft Lip Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Wake Forest University Health Sciences (Other); Boston Children's Hospital (Other); Massachusetts General Hospital (Other); Tufts Medical Center (Other); University of Bath (Other)
Responsible Party: Principal Investigator, Carroll Ann Trotman, Professor, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12250
Record Dates: First submitted 2018-02-15; First posted 2018-05-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cleft Palate; Cleft Lip
MeSH Terms: conditions — Cleft Palate; Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Static Images and Facial Videos (Other): 2D and 3D still and video images obtained from each patient before surgery.
  Interventions: Other: Static Images and Facial Videos

INTERVENTIONS:
Other: Static Images and Facial Videos — 2D and 3D still and video images obtained from each patient before surgery.

SUMMARY:
Using separate prospective cohorts of patients who have lip revision and lip repair surgery, the objective of this clinical trial is to both qualitatively and quantitatively assess how surgeons integrate the objective measures and visual aids of the Intervention with the systematic subjective assessment in order to determine decisions surgery.

DETAILED DESCRIPTION:
The standard-of-care to evaluate patients for lip revision surgery relies on a subjective assessment by the surgeon of the static face. The important role of function or movement generally has been given far less consideration mainly because of the challenges faced by surgeons (e.g., the amount/quality of the tissue available to alter movement). Presently, even when surgeons do attempt to assess function, they do so in a subjective manner because there are no quantitative/visual aids to incorporate functional assessment into their treatment planning and decisions regarding lip surgery.

The Intervention approach proposed here has been refined sufficiently with surgeon feedback to allow surgeons to broaden their "vista" of the patients' 'movement and form' problems. Potentially, having identified a movement/form problem(s), surgeons could contemplate what needs to be done to improve patient specific problem(s). Importantly, pilot studies demonstrated that the Intervention had a definite impact on surgeons' decisions for lip revision: Surgeons substantially, but variably, changed their problem list and treatment planning goals. Thus, a goal of this study is to collect surgical outcome data which will be used primarily to monitor adverse events but also will provide preliminary information on improvement in patient outcomes (facial form and movement) when surgeons use the Intervention. In addition, given that revision surgery is very common after the primary lip repair, it is important to understand surgeons' decision-making with the use of the Intervention, to determine surgeons' goals and expectations for primary lip repair surgery, and to understand the surgical limitations that may lead to subsequent revision surgery.

ELIGIBILITY:
Inclusion Criteria (Lip Revision):

* Age 4 to 21 years
* Presence of a previously repaired unilateral or bilateral cleft lip and palate with a complete cleft of the primary palate and at least a partial or complete cleft of the secondary palate
* The professional clinical recommendation by the craniofacial plastic surgeon for a full or partial thickness lip revision

Exclusion Criteria (Lip Revision):

* Lip revision surgery within the past two years
* A diagnosis of a craniofacial anomaly other than cleft lip (and palate)
* A medical history of collagen vascular disease, or systemic neurologic impairment
* Mental, visual, or hearing impairment to the extent that comprehension or ability to perform tests associated with the collection of the imaging data is hampered

Inclusion Criteria (Lip Repair)

* Age birth to 8 months
* Presence of an unrepaired unilateral or bilateral cleft lip and palate with a complete cleft of the primary palate and at least a partial or complete cleft of the secondary palate

Exclusion Criteria (Lip Repair)

* A diagnosis of a craniofacial anomaly other than cleft lip (and palate)
* A medical diagnosis of collagen vascular disease, and systemic neurologic impairment
* Mental, visual, or hearing impairment to the extent that the infant's ability to perform tests associated with the collection of the imaging data is hampered

Ages: 0 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Surgeon-raters' decision making in lip revision | Through study completion, an average of 2 years
  Outcomes are based on transcribing the In-Depth-Interviews (IDIs) that will be conducted with the surgeon-raters; coding the transcript with an a priori structure in mind (using the interview format as a starting point) but then using Grounded Theory to guide further coding in order to capitalize on themes that emerge that may not conform to the interview format. Themes will be developed (from the interview format and/or the emergent themes) that we will group by frequency as well as to their relevance to hypothesis generation as to how surgeon-raters might learn about and integrate patient data over time.
Surgeon-raters' decision making in primary lip repair | Through study completion, an average of 2 years
  Outcomes are based on transcribing the IDIs that will be conducted with the surgeon-raters; coding the transcript with an a priori structure in mind (using the interview format as a starting point) but then using Grounded Theory to guide further coding in order to capitalize on themes that emerge that may not conform to the structured interview format. Themes will be developed (from the interview format and/or the emergent themes) that we will group by frequency as well as to their relevance to hypothesis generation as to how surgeon-raters might learn about and integrate patient data over time.
  This thematic and frequency analysis will be conducted after the SAFS Intervention is conducted with the surgeons for those patients who are in need of lip revision surgery to address objective 1, as well as after the SAFS Intervention is conducted with the surgeons for those patients in need of primary lip repair surgery to address objective 2.

SECONDARY OUTCOMES:
The quantitative assessment of the extent to which the SAFS changes surgeon-raters' problem list and treatment planning goals for lip revision. | Through study completion, an average of 2 years
  Nominal outcome of the effect of the SAFS on surgeon-raters' treatment plans/goals in terms of whether the surgeon-rater changes his problem list and goals for lip revision.
The quantitative assessment of the extent to which the SAFS changes surgeons' problem list and treatment planning goals for primary lip repair. | Through study completion, an average of 2 years
  Nominal outcome of the effect of the SAFS on surgeon-raters' treatment plans/goals in terms of whether and how much the surgeon-rater changes his problem list and goals for primary lip repair.
The quantitative assessment of the extent to which the SAFS changes surgeon-raters' problem list and treatment planning goals for lip revision as a function of surgical expertise. | Through study completion, an average of 2 years
  Nominal outcome of the effect of the SAFS on surgeon-raters' treatment plans/goals in terms of whether the surgeon-rater changes his problem list and goals for lip revision based on the length of surgical experience (in years) of treating patients with cleft lip and palate.

CONTACTS AND LOCATIONS:
Overall Officials: Carroll Ann Trotman, Principal Investigator — Tufts University School of Dental Medicine
Locations (2):
- United States (2):
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No